CLINICAL TRIAL: NCT02500004
Title: Brown Adipose Tissue Activity and Energy Metabolism in Cachexia Induced by Cancer or Chronic Disease
Brief Title: Brown Adipose Tissue Activity and Energy Metabolism in Cachexia
Acronym: BAT-Cachexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 142071; NL51402.068.14 (Other: CCMO)
Record Dates: First submitted 2015-06-24; First posted 2015-07-16 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2016-03

CONDITIONS: Cachexia; Neoplasms; Pulmonary Disease, Chronic Obstructive; Pancreatic Neoplasms
MeSH Terms: conditions — Cachexia; Neoplasms; Pulmonary Disease, Chronic Obstructive; Pancreatic Neoplasms | interventions — Blood Specimen Collection; Calorimetry, Indirect; Accelerometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cachectic pancreatic cancer (Active Comparator): Cachectic patients with pancreatic cancer
  BAT activity: 18F-FDG PET-MRI-imaging. Body composition: DXA scanning, D2O and MRI. Inflammatory and metabolic profile of adipose tissue: abdominal subcutaneous adipose tissue biopsy.
  Systemic inflammatory profile: blood sampling. Resting metabolic rate: indirect calorimetry. Physical activity level: accelerometry. Total daily energy expenditure: double-labeled water.
  Interventions: Radiation: 18F-FDG PET-MRI-imaging; Radiation: DXA scanning; Procedure: Abdominal subcutaneous adipose tissue biopsy; Procedure: Blood sampling; Other: Indirect calorimetry; Device: Accelerometry; Other: Double-labeled water
- Cachectic NSCLC (Active Comparator): Cachectic patients with non-small cell lung cancer
  BAT activity: 18F-FDG PET-MRI-imaging. Body composition: DXA scanning, D2O and MRI. Inflammatory and metabolic profile of adipose tissue: abdominal subcutaneous adipose tissue biopsy.
  Systemic inflammatory profile: blood sampling. Resting metabolic rate: indirect calorimetry. Physical activity level: accelerometry. Total daily energy expenditure: double-labeled water.
  Interventions: Radiation: 18F-FDG PET-MRI-imaging; Radiation: DXA scanning; Procedure: Abdominal subcutaneous adipose tissue biopsy; Procedure: Blood sampling; Other: Indirect calorimetry; Device: Accelerometry; Other: Double-labeled water
- Cachectic COPD (Active Comparator): Cachectic COPD patients.
  BAT activity: 18F-FDG PET-MRI-imaging. Body composition: DXA scanning, D2O and MRI. Inflammatory and metabolic profile of adipose tissue: abdominal subcutaneous adipose tissue biopsy.
  Systemic inflammatory profile: blood sampling. Resting metabolic rate: indirect calorimetry. Physical activity level: accelerometry. Total daily energy expenditure: double-labeled water.
  Interventions: Radiation: 18F-FDG PET-MRI-imaging; Radiation: DXA scanning; Procedure: Abdominal subcutaneous adipose tissue biopsy; Procedure: Blood sampling; Other: Indirect calorimetry; Device: Accelerometry; Other: Double-labeled water
- Non-cachectic COPD (Active Comparator): Non-cachectic COPD patients.
  BAT activity: 18F-FDG PET-MRI-imaging. Body composition: DXA scanning, D2O and MRI. Inflammatory and metabolic profile of adipose tissue: abdominal subcutaneous adipose tissue biopsy.
  Systemic inflammatory profile: blood sampling. Resting metabolic rate: indirect calorimetry. Physical activity level: accelerometry. Total daily energy expenditure: double-labeled water.
  Interventions: Radiation: 18F-FDG PET-MRI-imaging; Radiation: DXA scanning; Procedure: Abdominal subcutaneous adipose tissue biopsy; Procedure: Blood sampling; Other: Indirect calorimetry; Device: Accelerometry; Other: Double-labeled water
- Healthy individuals (Other): BAT activity: 18F-FDG PET-MRI-imaging. Body composition: DXA scanning, D2O and MRI. Inflammatory and metabolic profile of adipose tissue: abdominal subcutaneous adipose tissue biopsy.
  Systemic inflammatory profile: blood sampling. Resting metabolic rate: indirect calorimetry. Physical activity level: accelerometry. Total daily energy expenditure: double-labeled water.
  Interventions: Radiation: 18F-FDG PET-MRI-imaging; Radiation: DXA scanning; Procedure: Abdominal subcutaneous adipose tissue biopsy; Procedure: Blood sampling; Other: Indirect calorimetry; Device: Accelerometry; Other: Double-labeled water

INTERVENTIONS:
Radiation: 18F-FDG PET-MRI-imaging — BAT activity: 18F-FDG PET-MRI-imaging.
Radiation: DXA scanning — Body composition: DXA scanning, D2O and MRI.
Procedure: Abdominal subcutaneous adipose tissue biopsy — Inflammatory and metabolic profile of adipose tissue: abdominal subcutaneous adipose tissue biopsy.
Procedure: Blood sampling — Systemic inflammatory profile: blood sampling.
Other: Indirect calorimetry — Resting metabolic rate: indirect calorimetry.
Device: Accelerometry — Physical activity level: accelerometry.
Other: Double-labeled water — Body composition: DXA scanning, D2O and MRI. Total daily energy expenditure: double-labeled water.

SUMMARY:
To study BAT activity and energy metabolism in patients with cachexia induced by cancer or chronic disease.

DETAILED DESCRIPTION:
This is a prospective, cross-sectional study to determine BAT activity in cachectic patients with pancreatic or non-small cell lung cancer, and in cachectic patients with chronic obstructive pulmonary disease (COPD), and compare results with healthy individuals and non-cachectic COPD patients, matched for age and BMI.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cancer patients, or NSCLC cancer patients, or COPD patients
* The diagnostic criterion for cachexia is unintentional weight loss more than 5% over the past 6 months or more than 2% in individuals with a body-mass index < 20 kg/m2 and muscle wasting assessed by DXA;
* Age ≥ 30 years;
* Gender: male and female;
* Caucasians.

Exclusion Criteria:

* Uncontrolled Diabetes Mellitus;
* Patients with severe clotting disorder;
* Patients with an active second malignancy;
* Psychological unstable persons presumed unfit to perform the measurements, including claustrophobia;
* Persons unable to lie or sit still for 1-2 hours;
* Oxygen therapy;
* Pregnant subjects;Subjects unable to undergo MRI (e.g. pacemaker; neurostimulator; implantable cardioverter-defibrillator (ICD) or leads; Foley bladder catheter; medication pump; cochlear or hearing implant; tattoos or other items that cannot be removed and include metal parts (for instance from operations in the past); metal splinter in the eye; vascular clips; denture, which contains magnets);
* Subjects that received high doses of radiotherapeutic radiation of the neck and/or upper chest in their medical history;
* Persons that received cervical or thoracic sympathectomy or have a nerve dysfunction which is likely to influence sympathetic nerves;
* The use of medication that influences the sympathetic nerve system: ß-blockers, α-blockers, central anti-hypertensives, certain anti-depression drugs (MAO inhibitors, tricyclic anti-depressives), reserpine, cocaine, calciumblockers, labetalol, and certain tranquillizers (fenothiazines).

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Brown adipose tissue (BAT) activity measured by PET(-MRI) | participants will be followed for 2 weeks
  The main endpoint of this study is BAT volume and intensity of activity in Standard Uptake Value (SUV) in the presence of cancer cachexia, COPD cachexia, and compared to non-cachectic COPD patients and healthy individuals, as assessed by 18F-fluoro-deoxyglucose (18F-FDG) PET-MRI scanning.

SECONDARY OUTCOMES:
Total energy metabolism measured by resting energy expenditure (REE) and doubly labeled water | participants will be followed for 2 weeks
Resting metabolic rate measured by REE | participants will be followed for 2 weeks
Metabolic gene expression in WAT measured by biopsy of subcutaneous fat | participants will be followed for 2 weeks
Systemic inflammatory status measured in blood | participants will be followed for 2 weeks
Fat tissue mass measured by MRI, DXA, and doubly labeled water | participants will be followed for 2 weeks
  Detailed body composition phenotyping of cachexia by (PET-)MRI to compare with commonly applied clinical measures (D2O and DXA)
Hormonal status measured in blood | participants will be followed for 2 weeks
Lean tissue mass measured by MRI, DXA, and doubly labeled water | participants will be followed for 2 weeks
  Detailed body composition phenotyping of cachexia by (PET-)MRI to compare with commonly applied clinical measures (D2O and DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Schols, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht UMC+, Maastricht, Netherlands

REFERENCES:
- [Derived] Sanders K, Klooster K, Vanfleteren LEGW, Plasqui G, Dingemans AM, Slebos DJ, Schols AMWJ. Effect of Bronchoscopic Lung Volume Reduction in Advanced Emphysema on Energy Balance Regulation. Respiration. 2021 Feb 5:1-8. doi: 10.1159/000511920. Online ahead of print. PMID 33550302